CLINICAL TRIAL: NCT04855383
Title: The Effect of Intramuscular Injection of Triple Doses of Human Chorionic Gonadotropin in Frozen Embryo Transfer Cycles
Brief Title: Intramuscular Injection of Human Chorionic Gonadotropin in Frozen Embryo Transfer Cycles
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Royan Institute (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FET-HCG
Record Dates: First submitted 2021-04-18; First posted 2021-04-22 (Actual); Last update posted 2024-01-05 (Actual); Status verified 2024-01

CONDITIONS: Embryo Implantation
Keywords: Human chorionic gonadotropin; frozen embryo transfer; infertility; assisted reproduction technology; estrogen/ progesterone replacement cycles
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The group of frozen embryo transfer with intramuscular injection of human chorionic gonadotropin. (Experimental): In this group, endometrial preparation for embryo transfer will be through the standard protocol using a gonadotropin-releasing hormone agonist. Patients receive 5,000 IU of human chorionic gonadotropin by intramuscular injection, 72 hours before embryo transfer, on the day of embryo transfer, and 72 hours after embryo transfer.
  Interventions: Drug: The effect of intramuscular injection of triple doses of human chorionic gonadotropin in frozen embryo transfer cycles
- The group of frozen embryo transfer without intramuscular injection of human chorionic gonadotropin. (No Intervention): In this group, endometrial preparation for embryo transfer will be through the standard protocol using a gonadotropin-releasing hormone agonist. Embryo transfer will be done without human chorionic gonadotropin intramuscular injection.

INTERVENTIONS:
Drug: The effect of intramuscular injection of triple doses of human chorionic gonadotropin in frozen embryo transfer cycles — Patients receive 5,000 IU of human chorionic gonadotropin by intramuscular injection, 72 hours before embryo transfer, on the day of embryo transfer, and 72 hours after embryo transfer.
  Other Names: The effect of intramuscular injection of triple doses of human chorionic gonadotropin on embryo implantation
  Arms: The group of frozen embryo transfer with intramuscular injection of human chorionic gonadotropin.

SUMMARY:
This study is a randomized controlled clinical trial to compare the pregnancy outcomes of infertile women with frozen embryo transfer. The study population in frozen embryo transfer cycles receive three doses of human chorionic gonadotropin (HCG) to recognize the effectiveness of HCG on pregnancy outcomes in Reproductive Biomedicine Research Center, Royan institute, Tehran Iran.

DETAILED DESCRIPTION:
During implantation, the biochemical crosstalk between the endometrium and embryo has a very important role. The endometrium secrets cytokines and growth factors that modulate embryonic differentiation and early development. One of the important molecular messages between the embryo and endometrium is human chorionic gonadotropin (HCG). HCG is expressed by the blastocyst before the implantation, while increasingly produced after implantation by the syncytiotrophoblast. In order to study the direct effect of HCG on the endometrium at implantation, this randomized, controlled clinical trial evaluated whether HCG supplementation would be beneficial for pregnancy outcomes of cryopreserved-thawed embryo transfer with estrogen/ progesterone replacement cycles at Royan Institute.

Block randomization method is designed by epidemiologist using STATA software version 13 and the number of blocks considered is 6. The random allocation list for patients is solely available to the epidemiologist. In order to hide the random allocation process, a total of 200 envelopes are prepared, and only the methodologist has been aware of table of random numbers. When the doctor declared the patient's eligibility, the methodologist provided the doctor with the envelope. The group will be selected and based on the type of group mentioned in the envelope.

ELIGIBILITY:
Inclusion Criteria:

* Infertile women candidates for frozen embryo transfer
* Age 20-40 years
* Body Mass Index under than 30 Kg/m2
* Having at least three good quality embryos

Exclusion Criteria:

* Women with hematologic and autoimmune disorders
* Couples with chromosomal and genetic abnormalities
* Women with uterine anomalies
* Women with uterine and ovaries surgical history
* Women with endometriosis and adenomyosis
* Women with hydrosalpinx
* Women with uterine fibroids
* Women with history of recurrent abortion or recurrent implantation failure
* Severe male factor infertility (azoospermia)
* Embryo donation cycle
* Endometrial thickness less than 8 millimeter on the day of embryo transfer

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 200 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2022-08-22 (Actual); Study Completion 2023-06-20 (Actual)

PRIMARY OUTCOMES:
Rate of Implantation | 6 weeks after embryo transfer
  Implantation rate is the percentage of embryos which successfully undergo implantation compared to the number of embryos transferred in a given period.

CONTACTS AND LOCATIONS:
Overall Officials: Mehri Mashayekhi, M.D., Study Director — Department of Endocrinology and Female Infertility, ACECR, Tehran, Iran.; Azar Yahyaei, M.Sc., Principal Investigator — Department of Endocrinology and Female Infertility, ACECR, Tehran, Iran.
Locations (1):
- Royan Institute, Tehran, Iran

IPD SHARING:
Plan to Share IPD: Yes
After the publication of the article Available to the public. Scientific use by citing the source. Request via e-mail
Supporting Information: CSR
Time Frame: After the publication of the article
Access Criteria: Available to the public. Scientific use by citing the source.